CLINICAL TRIAL: NCT05223517
Title: Effect of Acupuncture for Chronic Pelvic Pain in Women: a Randomized Clinical Trial
Brief Title: Acupuncture for Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-135-KY-01
Record Dates: First submitted 2022-01-06; First posted 2022-02-04 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Acupuncture, Chronic Pelvic Pain, Woman
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupucnture (Experimental)
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — Hwato brand disposable acupuncture needles (size 0.30 × 40 mm and 0.30 × 75 mm) and adhesive pads will be used. Acupoints of Ciliao, Huiyang, Shenshu, Guanyuan, Shuidao, Sanyinjiao, Zusanli, Taixi, Hegu, and Taichong will be used for every participants. Those with sleep or mood disorders will also use acupoints of Shangyintang, Shenmen and Neiguan. Those with tenderness points on the abdominal wall will also use Ashi points no more than five.
  The needles will be inserted to 60-70mm in Ciliao and Huiyang, 6-10 mm in Shenmen and 10-20mm in other acupoints through adhesive pads. Needles will be lifted, thrusted and twirled gently for 3 times (except for Ciliao) to achieve deqi sensation and manipulated every ten minutes during 20-minute maintenance in prone and supine position respectively.
  Participants receive acupuncture treatment three times a week in the first four weeks and twice a week in the last four weeks.
  Arms: Acupucnture
Device: Sham Acupuncture — Hwato brand disposable placebo needles (with the handle identical to the needles in the acupuncture group and the body at a size 0.30 × 25 mm) and adhesive pads will be used. Acupoints of Ciliao, Huiyang, Shenshu, Guanyuan, Shuidao, Sanyinjiao, Zusanli, Taixi, Hegu, and Taichong will be used for every participants. Those with sleep or mood disorders will also use acupoints of Shangyintang, Shenmen and Neiguan. Those with tenderness points on the abdominal wall will also use Ashi points no more than five.
  The needles will be inserted into adhesive pads without skin penetration. Needles will be lifted, thrusted and twirled gently for 3 times to mimic real acupuncture. No manipulation will be conducted during 20-minute maintenance in prone and supine position respectively.
  Participants receive sham acupuncture treatment three times a week in the first four weeks and twice a week in the last four weeks.
  Arms: Sham Acupuncture

SUMMARY:
The aim of the study is to assess the effects and safety of acupuncture for moderate to severe chronic pelvic pain in women.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 50.
* Chronic pelvic pain (with or without dysmenorrhoea or dyspareunia) of at least 6 months duration.
* Having not used medications, other than rescue medicine, or therapies for chronic pelvic pain for at least 4 weeks before randomization, and consenting not to use throughout the process of the research.
* Completing Weekly Pain Diary for at least three week during the four-week run-in period, and at least two of the worst pain scoring ≥4 on the Numeric Rating Scale.
* Volunteering to participate the trial and signing written informed consent.

Exclusion Criteria:

* Cyclical chronic pelvic pain, such as only with dysmenorrhea.
* Endometriosis.
* Adenomyosis.
* Complex ovarian cyst.
* Accessory cyst >5cm.
* Uterine fibroids >5cm.
* Malignant disease.
* Anterior sacral neurectomy or uterine sacral nerve ablation before or scheduled in the next 6 month.
* Irritable bowel syndrome.
* Symptomatic urinary tract infection.
* Acute pelvic inflammation.
* Uncontrolled vaginitis.
* Lactation period, pregnancy, or fetation planned in the next 6 months.
* Sever disorders in heart, lung, brain, liver, kidney and hematopoietic system, or obvious psychiatric or cognitive dysfunction.
* Poor adherence.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-03-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with at least 50% reduction of numerical rating scale (NRS) score on average pain. | Weeks 5-8
  Participants will rate their average chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of the four weeks.

SECONDARY OUTCOMES:
Proportion of participants with at least 50% reduction of numerical rating scale (NRS) score on average pain. | Weeks 1-4, 9-12, 13-16, 17-20.
  Participants will rate their average chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of the four weeks.
Proportion of participants with at least 50% reduction of numerical rating scale (NRS) score on the worst pain. | Weeks 1-4, 5-8, 9-12, 13-16, 17-20.
  Participants will rate their worst chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the four weeks will be taken as final NRS score on the worst pain.
The change from baseline in the numerical rating scale (NRS) score on average pain. | Weeks 1-4, 5-8, 9-12, 13-16, 17-20.
  Participants will rate their average chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of the four weeks.
The change from baseline in the numerical rating scale (NRS) score on the worst pain. | Weeks 1-4, 5-8, 9-12, 13-16, 17-20.
  Participants will rate their worst chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the four weeks will be taken as final NRS score on the worst pain.
Proportion of participants with at least 30% reduction of numerical rating scale (NRS) score on average pain. | Weeks 1-4, 5-8, 9-12, 13-16, 17-20.
  Participants will rate their average chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The final NRS score on average pain is defined as the mean of the average pain scores of the four weeks.
Proportion of participants with at least 30% reduction of numerical rating scale (NRS) score on the worst pain. | Weeks 1-4, 5-8, 9-12, 13-16, 17-20.
  Participants will rate their worst chronic pelvic pain each week on a 0-10 NRS scale, where 0 refers to no pain and 10 refers to the worst pain imaginable. The highest worst pain score of the four weeks will be taken as final NRS score on the worst pain.
The change from baseline in the interferes score of Brief Pain Inventory (BPI) short form. | Weeks 4, 8, 12, 16, 20
  The Brief Pain Inventory (BPI) short form assesses the degree to which the chronic pelvic pain interferes with activities over the prior week in terms of general activity, mood, walking ability, normal work (including housework), relations with other people, sleep and enjoyment of life using a 0- to 10-point scale (0 [Does not interfere] to 10 [Completely interferes]).
The proportion of participants rates their overall improvement as "very much improved" or "much improved" based on the Patient Global Impression-Change (PGI-C) . | Weeks 8 and 20
  The Patient Global Impression-Change (PGI-C) is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse" or "very much worse".
The change from baseline in the Female Sexual Function Index (FSFI) score. | Weeks 8 and 20
  The Female Sexual Function Index (FSFI) is a 19-item self-report inventory designed to assess female sexual function, which comprises six domains of desire, arousal, lubrication, orgasm, satisfaction, and pain.
The change from baseline in the total and sub scores of Hospital Anxiety and Depression Scale (HADS). | Weeks 4, 8 and 20
  Hospital Anxiety and Depression Scale (HADS) consists of 14 items, divided into two 7 item subscales to reflect a state of generalized anxiety and the depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence).
The change from baseline in the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire. | Weeks 4, 8 and 20
  EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire is used to measure health-related quality of life. It consists of five questions about mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, and a visual analogue scale on the general health state during the day.

OTHER OUTCOMES:
Expectance assessment | Baseline
  Participants will be asked what do you think the condition of chronic pelvic pain will be in two month?
Assessment of belief in acupuncture | Baseline, week 4, week 8
  Participants will be asked do you think acupuncture will help to treat your chronic pelvic pain.
Blinding assessment | Within 5 minutes after either treatment in week 8
  Participants will be ask do you think you have received traditional acupuncture in the past 8 weeks.
Adherence assessment | Weeks 1-8
  Adherence will be assessment via counting treatment sessions. Those complete over 80% treatment sessions will be defined as of good adherence.
Proportion of participants using rescue medicine. | Through study completion, an average of 3 years
Proportion of participants using concomitant medicine or therapy that might impact chronic pelvic pain. | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with publication until six months after publication.
  Formal request should be sent to puzhisun@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until until six months after publication.
Access Criteria: Formal request should be sent to puzhisun@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.